CLINICAL TRIAL: NCT05487443
Title: An Open, Single-arm Prospective Clinical Study Evaluating the Efficacy of Systemic Venous Gemcitabine-based Chemotherapy Combined With Immunocheckpoint Inhibitors in First-line Treatment of Advanced Biliary Malignancies
Brief Title: The Efficacy of Chemotherapy Combined With Immunocheckpoint Inhibitors in Advanced Biliary Malignancies
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20211216
Record Dates: First submitted 2021-12-27; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2021-12

CONDITIONS: Gemcitabine; Biliary Tract Cancer; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy combined with immunotherapy (Experimental): Gemcitabine-based chemotherapy regimen combined with immunocheckpoint inhibitors for first-line treatment of advanced biliary malignancies
  Interventions: Drug: Gemcitabine-based chemotherapy regimen combined with immunocheckpoint inhibitors

INTERVENTIONS:
Drug: Gemcitabine-based chemotherapy regimen combined with immunocheckpoint inhibitors — Gemcitabine-based chemotherapy regimen combined with immunocheckpoint inhibitors for first-line treatment of advanced biliary malignancies

SUMMARY:
To the patient of terminal biliary malignancy tumor, how should the patient's treatment plan choose ? To address this problem, this study intends to analyze systemic venous gemcitabine-based chemotherapy regimen combined with immune checkpoint inhibitors in patients with advanced BTC, to evaluate the long-term efficacy and toxicity of patients, and to search for predictable biomarkers. In order to clarify the advantages and disadvantages of intravenous chemotherapy combined with immunotherapy for patients with advanced biliary malignancy, provide certain basis for clinical work, and then select the most suitable treatment plan for patients according to the different characteristics of individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Non-bedridden male or female, aged ≥18 years and ≤80 years. Adopts the surgery of Chinese medical association branch of biliary surgery group released the diagnosis and treatment of the bile duct carcinoma surgery expert consensus on biliary tract tumor diagnosis standard, refer to biliary lining after epithelial malignant tumors, including intrahepatic bile duct carcinoma, liver bile duct carcinoma, distal bile duct carcinoma and portal vein gallbladder, or postoperative pathology biopsy for biliary tumor, Staging was performed according to the Joint Council on Cancer (AJCC) TNM version 8.
* the ECOG score of 0 to 2 points.
* the histologic diagnosis of unresectable locally advanced, recurrent and/or metastatic malignant tumor, biliary pathology for adenocarcinoma, untreated or always neoadjuvant therapy/adjuvant therapy over time to relapse time > 6 months.
* not intentional, liver, brain, kidney and other important organ dysfunction and bleeding tendency; No history of blood diseases; Cardiac insufficiency, chest pain (medically uncontrollable). No myocardial infarction occurred during the 12 months prior to the study.
* the subjects baseline blood routine and biochemical indexes in accordance with the following standards: 80 g/L or higher hemoglobin; Neutrophil absolute count (ANC) ≥1.5×109/L; Platelet ≥100×109/L; ALT, AST≤2.5 times the normal upper limit; ALP≤2.5 times normal upper limit value; Serum total bilirubin <1.5 times normal upper limit; Serum creatinine <1 times normal upper limit; Serum albumin ≥30g/L.
* there are measurable evaluation target lesions according to the RECIST criteria.

Exclusion Criteria:

* Younger than 18 or more than 76 years old (inclusive); Or poor general condition, ECOG score > 2.
* participated in other clinical trials.
* a blood coagulation dysfunction or history or severe clinical haematology (activities) heart disease, such as symptomatic coronary heart disease (CHD), New York heart association (NYHA) class II or more severe congestive heart failure or severe arrhythmia, drug intervention or within the past 12 months has a history of myocardial infarction.
* patients with past history has obvious liver and kidney function is not complete.
* Pregnancy and lactation women, women of childbearing age in the baseline period pregnancy test positive pregnancy test subjects or not. Menopausal women must be in menopause for at least 12 months before pregnancy is considered impossible.
* multi-source patients with carcinoma and repetition, or brain or meningeal metastasis. All landowners have uncontrolled seizures, central nervous system disease or a history of mental disorders, t

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 1 month

SECONDARY OUTCOMES:
Overall survival (OS) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided